CLINICAL TRIAL: NCT06246448
Title: Robotic-assisted Contra Open Resection for Suspected or Confirmed Gallbladder Cancer - An International, Multi-centre, Single Blinded, Randomized Controlled Superiority Trial
Brief Title: Robotic-assisted Contra Open Resection for Suspected or Confirmed Gallbladder Cancer (ROBOCOP)
Acronym: ROBOCOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: University Hospital, Linkoeping (Other); Sahlgrenska University Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Christian Sturesson, Associate professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CS001
Record Dates: First submitted 2024-01-22; First posted 2024-02-07 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Gall Bladder Cancer
MeSH Terms: conditions — Gallbladder Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robotic-assisted radical cholecystectomy (Experimental)
  Interventions: Procedure: Robotic-assisted radical cholecystectomy
- Open radical cholecystectomy (Active Comparator)
  Interventions: Procedure: Open radical cholecystectomy

INTERVENTIONS:
Procedure: Robotic-assisted radical cholecystectomy — Procedure will be performed robotic-assisted
  Arms: Robotic-assisted radical cholecystectomy
Procedure: Open radical cholecystectomy — Procedure will be open
  Arms: Open radical cholecystectomy

SUMMARY:
The Robocop trial is an international multi-centre, single blinded, randomized controlled superiority trial conducted in centres experienced in robotic-assisted liver surgery. Eligible patients for radical cholecystectomy will be randomized in a 1:1 ratio to undergo robotic-assisted or open resection within an enhanced recovery setting.

The primary endpoint is time to functional recovery. Secondary endpoints include length of hospital stay, resection margin, number of retrieved lymph nodes, postoperative complications, quality of life, abdominal wall complaints and direct and indirect costs.

DETAILED DESCRIPTION:
Robotic-assisted surgery is hypothesised to reduce time to functional recovery by 2 days compared with open surgery. With a power of 80% and alpha of 0.05, the sample size needed in each arm to test superiority is 35 patients. With an expected 25% drop-out rate, 47 patients will be randomized in each group, with a total of 94 patients to be randomized in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient with radiologically suspected or confirmed (≥T1b) incidental gallbladder cancer after cholecystectomy with an indication of radical cholecystectomy, without the need for resection of extrahepatic bile ducts, as decided at a multidisciplinary team conference.
* Patient sufficiently fit to undergo radical cholecystectomy according to surgeon and anaesthesiologist.

Exclusion Criteria:

* Previous extensive surgery in the upper abdomen (for example open liver surgery)
* Pregnancy
* Intraoperative findings of dissemination (patient is then excluded after randomization)
* Intraoperative findings of the need to perform resection of extrahepatic bile ducts (patient is then excluded after randomization).
* Intraoperative findings leading to a simple cholecystectomy only (patient is then excluded after randomization)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Time to functional recovery | Days from operation
  As defined as: 1. has adequate pain control with oral analgesics only (NRS<5) 2. is independently mobile at the preoperative level 3. is able to maintain sufficient oral caloric intake (minimum of 50% required calories) 4. has no need for intravenous fluid administration 5. has no clinical signs of infection or infection treated with peroral antibiotics only

SECONDARY OUTCOMES:
Number of retrieved lymph nodes | Within 6 weeks after surgery
  As reported by pathologists
Length of hospital stay | Days
  Time from operation until hospital discharge (days)
Post-operative complications | Within 90 days from surgery
  Classified according to Clavien-Dindo
Quality of life of patients | 1 year
  Using quality of life formulaire EORTC QLQ-C30
Total cost | 1 year
  Direct and indirect cost measured in euros
Abdominal wall complaints | 1 year
  Using the ventral hernia pain questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Christian Sturesson, PhD, Principal Investigator — Region Stockholm, Stockholm, Sweden
Locations (1):
- Region Stockholm, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wallgren H, Gilg S, Ansorge C, Sparrelid E, Sturesson C. Initial experience with robotic-assisted resection for suspected or confirmed gallbladder cancer - comparison with open technique in a single centre retrospective observational cohort study. Scand J Gastroenterol. 2025 Jul 7:1-6. doi: 10.1080/00365521.2025.2525902. Online ahead of print. PMID 40621784